CLINICAL TRIAL: NCT03998761
Title: Micronized Progesterone Versus Micronized Progesterone Plus Dydrogesterone for Luteal Phase Support in Frozen - Thawed Transfer: a Prospective Cohort Study
Brief Title: Progesterone Versus Progesterone Plus Dydrogesterone in FET
Acronym: MiDRONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS/BVMĐ/19/06
Record Dates: First submitted 2019-06-17; First posted 2019-06-26 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Infertility
Keywords: FET; Micronized Progesterone; Dydrogesterone
MeSH Terms: conditions — Infertility | interventions — Progesterone; Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Micronized progesterone (Active Comparator): Patients will receive micronized progesterone (Cyclogest® 400mg; Actavis) at the dose of 400mg twice daily (morning and evening).
  Interventions: Drug: Micronized Progesterone
- Micronized progesterone plus dydrogesterone (Active Comparator): Patients will receive micronized progesterone (Cyclogest® 400mg; Actavis) at the dose of 400mg twice daily (morning and evening) plus dydrogesterone (Duphaston® 10mg, Abbott) at the dose of 10mg twice daily (morning and evening).
  Interventions: Drug: Micronized progesterone plus dydrogesterone

INTERVENTIONS:
Drug: Micronized Progesterone — Progesterone will be started when endometrial thickness reached 8 mm or more. Patients will receive micronized progesterone (Cyclogest® 400mg; Actavis) at the dose of 400mg twice daily (morning and evening). A maximum of 2 embryos will be thawed on the day of embryo transfer, which is four days or six days after the start of progesterone depending on day-3 or day-5 embryo transfer. After thawing, surviving embryos will be transferred into the uterus under ultrasound guidance. Estradiol and progesterone will be continued until the day of pregnancy test. If the pregnancy test is positive, the patients will continue to use 800 mg micronized progesterone until 7 weeks of gestation.
  Other Names: Cyclogest 400mg
  Arms: Micronized progesterone
Drug: Micronized progesterone plus dydrogesterone — Progesterone will be started when endometrial thickness reached 8 mm or more. Patients will receive micronized progesterone (Cyclogest® 400mg; Actavis) at the dose of 400mg twice daily (morning and evening) plus dydrogesterone (Duphaston® 10mg, Abbott) at the dose of 10mg twice daily (morning and evening). A maximum of 2 embryos will be thawed on the day of embryo transfer, which is four days or six days after the start of progesterone depending on day-3 or day-5 embryo transfer. After thawing, surviving embryos will be transferred into the uterus under ultrasound guidance. Estradiol and progesterone will be continued until the day of pregnancy test. If the pregnancy test is positive, the patients will continue to use 800 mg micronized progesterone plus 20 mg dydrogestetrone until 7 weeks of gestation.
  Other Names: Cyclogest 400 mg + Duphaston 10 mg
  Arms: Micronized progesterone plus dydrogesterone

SUMMARY:
Frozen embryo transfer (FET) has been increasing important in IVF. Progesterone is essential for the endometrial secretory transformation, establishment and maintenance of pregnancy. In FET, as there is neither corpus luteum nor the support of hCG, the role of progesterone is even more important to ensure a sufficient luteal phase support.

Vaginal progesterone has been the most common preparation for luteal support in fresh embryo transfer during IVF because of their ease of use and comparable effectiveness compared to intramuscular progesterone. Recently, there was evidence of the considerable variation in uptake, absorption and metabolism of intra-vaginal micronized progesterone. Dydrogesterone alone has described to have similar effectiveness, safety and tolerability prolfiles for luteal phase support compared to vaginal progesterone in luteal phase support for fresh embryo transfer. This prospective study compares the effectiveness of micronized progesterone versus micronized progesterone plus dydrogesterone for luteal phase support in FET.

DETAILED DESCRIPTION:
All patients undergoing FET will receive oral estradiol valerate (Valiera®; Laboratories Recalcine) 8 mg/day from the second or third day of menses for 6 days. Endometrial thickness will be monitored from day six onwards. From day 8-9 of menses, the estradiol dose could be adjusted from 8mg/day to 16mg/day according the development of the endometrium. Progesterone will be started when endometrial thickness reached 8 mm or more. In the first four months, all the patients will be treated with micronized progesterone. In five months later, the intervention will be changed to micronized progesterone plus dydrogesterone. In the second group of patients, the duration of study will be extended for one month due to the Lunar New Year holiday.

Group 1: Micronized progesterone Patients will receive micronized progesterone (Cyclogest® 400mg; Actavis) at the dose of 400mg twice daily (morning and evening).

Group 2: Micronized progesterone plus dydrogesterone Patients will receive micronized progesterone (Cyclogest® 400mg; Actavis) at the dose of 400mg twice daily (morning and evening) plus dydrogesterone (Duphaston 10mg) at the dose of 10mg twice daily (morning and evening).

In both group, on the day of starting progesterone, the dose of estradiol will be decreased to 8mg/day. A maximum of 2 embryos will be thawed on the day of embryo transfer, which is four days or six days after the start of progesterone depending on day-3 or day-5 embryo transfer. After thawing, surviving embryos will be transferred into the uterus under ultrasound guidance. Estradiol and progesterone will be continued until the day of pregnancy test. If the pregnancy test is positive, the patients will continue to use 800 mg micronized progesterone or 800 mg micronized progesterone plus 20 mg dydrogestetrone, until 7 weeks of gestation.

Blood samples will be obtained at day 4 after the use of progesterone. Serum progesterone will be measured. The blood tests will be taken in the morning, 2-3 h after the dydrogesterone and/or micronized progesterone application.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing frozen embryo transfer
* Endometrial prepared by exogenous hormonal regimen
* Permanent resident in Vietnam

Exclusion Criteria:

* Having > 2 embryo transfer attempts
* Having embryo(s) from donors cycles
* Having embryo(s) from IVM
* Having embryo(s) from PGT/PGS
* Having endometrial abnormalities: polyp, sub-mucosal fibroid, cesarean scar defects, endometrial hyperplasia, endometrial fluid accumulation, endometrial adhesion.
* Participating in another IVF study at the same time

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1364 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Live birth rate | At least 24 weeks of gestation up to the time of delivery
  The birth of at least one newborn after 24 weeks of gestation that exhibits any sign of life such as respiration, heartbeat, umbilical pulsation or movement of voluntary muscles (twin will be a single count).

SECONDARY OUTCOMES:
The luteal progesterone level | On day four of the progesterone application
  The progesterone level in serum on day four after the progesterone application
The length of luteal phase | On day sixteen of progesterone application
  Starting on the day of progesterone application and ending on the last day prior menses
Positive pregnancy test rate | On day sixteen of progesterone application
  Serum human chorionic gonadotropin level greater than 5 mIU/mL after the completion of the first transfer
Clinical pregnancy rate | At 7 weeks of gestation
  At least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity after the completion of the first transfer
Ongoing pregnancy rate | At 12 weeks' gestation
  Pregnancy with detectable heart rate at 12 weeks' gestation or beyond after the completion of the first transfer.
Implantation rate rate | At 3 weeks after embryo transferred
  The number of gestational sacs per number of embryos transferred after the completion of the first transfer.
Ectopic pregnancy rate | At 12 weeks of gestation
  A pregnancy in which implantation takes place outside the uterine cavity
Miscarriage rate | At 12 weeks of gestation
  Pregnancy loss at < 12 weeks
Multiple pregnancy rate | At 7 weeks' gestation
  Presence of more than one sac at early pregnancy ultrasound (6-8 weeks of gestation)
Gestational diabetes rate | At 24 weeks of gestation
  A type of diabetes that develop during pregnancy
Hypertensive disorder of pregnancy rate | From 20 weeks of gestation up to at birth
  Comprising pregnancy induced hypertension (PIH); pre-eclampsia (PET) and eclampsia
Antepartum haemorrhage rate | From 24 weeks of gestation up to at birth
  Defined as bleeding from or in to the genital tract, occurring from 24 weeks of pregnancy and prior to the birth of the baby, including placenta previa, placenta accreta and unexplained
Preterm delivery rate | At birth
  Defined as delivery at <24, <28, <32, <37 completed weeks
Birth weight (grams) of singletons and twins | At birth
  Weight of baby born (grams)
Low birth weight rate | At birth
  Weight of baby born < 2500 g at birth
Very low birth weight rate | At birth
  Weight of baby born < 1500 g at birth
High birth weight rate | At birth
  Weight of baby born >4000 gm at birth
Very high birth weight rate | At birth
  Weight of baby born > 4500 gm at birth
Congenital anomaly diagnosed at birth rate | At birth
  Any congenital anomalies detected in baby born
Venous thromboembolism (VTE) rate | At 7 weeks of gestation
  Including deep venous thrombosis and pulmonary embolism
Gastrointestinal disorders rate | At 7 weeks of gestation
  Including nausea, bloating, elevated liver enzymes
Nervous system disorders rate | At 7 weeks of gestation
  Including headache, dizziness
Vaginal discharge rate | At 7 weeks of gestation
  A fluid produced by glands in the vaginal wall and cervix that drains from the opening of the vagina
Vaginal discomfort rate | At 7 weeks of gestation
  Including the symptoms of pain, itching, burning and swelling of vagina and vulva
Vulvovaginal pruritus rate | At 7 weeks of gestation
  Itchiness of the vulva and vagina

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Study Chair — Hope Research Center
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Tan Binh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbosa MW, Silva LR, Navarro PA, Ferriani RA, Nastri CO, Martins WP. Dydrogesterone vs progesterone for luteal-phase support: systematic review and meta-analysis of randomized controlled trials. Ultrasound Obstet Gynecol. 2016 Aug;48(2):161-70. doi: 10.1002/uog.15814. Epub 2016 Jul 8. PMID 26577241
- [Background] Griesinger G, Blockeel C, Sukhikh GT, Patki A, Dhorepatil B, Yang DZ, Chen ZJ, Kahler E, Pexman-Fieth C, Tournaye H. Oral dydrogesterone versus intravaginal micronized progesterone gel for luteal phase support in IVF: a randomized clinical trial. Hum Reprod. 2018 Dec 1;33(12):2212-2221. doi: 10.1093/humrep/dey306. PMID 30304457
- [Background] Griesinger G, Blockeel C, Tournaye H. Oral dydrogesterone for luteal phase support in fresh in vitro fertilization cycles: a new standard? Fertil Steril. 2018 May;109(5):756-762. doi: 10.1016/j.fertnstert.2018.03.034. PMID 29778368
- [Background] Tournaye H, Sukhikh GT, Kahler E, Griesinger G. A Phase III randomized controlled trial comparing the efficacy, safety and tolerability of oral dydrogesterone versus micronized vaginal progesterone for luteal support in in vitro fertilization. Hum Reprod. 2017 May 1;32(5):1019-1027. doi: 10.1093/humrep/dex023. PMID 28333318
- [Background] Wang Y, He Y, Zhao X, Ji X, Hong Y, Wang Y, Zhu Q, Xu B, Sun Y. Crinone Gel for Luteal Phase Support in Frozen-Thawed Embryo Transfer Cycles: A Prospective Randomized Clinical Trial in the Chinese Population. PLoS One. 2015 Jul 29;10(7):e0133027. doi: 10.1371/journal.pone.0133027. eCollection 2015. PMID 26222435
- [Background] Wei D, Liu JY, Sun Y, Shi Y, Zhang B, Liu JQ, Tan J, Liang X, Cao Y, Wang Z, Qin Y, Zhao H, Zhou Y, Ren H, Hao G, Ling X, Zhao J, Zhang Y, Qi X, Zhang L, Deng X, Chen X, Zhu Y, Wang X, Tian LF, Lv Q, Ma X, Zhang H, Legro RS, Chen ZJ. Frozen versus fresh single blastocyst transfer in ovulatory women: a multicentre, randomised controlled trial. Lancet. 2019 Mar 30;393(10178):1310-1318. doi: 10.1016/S0140-6736(18)32843-5. Epub 2019 Feb 28. PMID 30827784
- [Background] Yanushpolsky E, Hurwitz S, Greenberg L, Racowsky C, Hornstein M. Crinone vaginal gel is equally effective and better tolerated than intramuscular progesterone for luteal phase support in in vitro fertilization-embryo transfer cycles: a prospective randomized study. Fertil Steril. 2010 Dec;94(7):2596-9. doi: 10.1016/j.fertnstert.2010.02.033. Epub 2010 Mar 27. PMID 20347079
- [Background] Labarta E, Mariani G, Holtmann N, Celada P, Remohi J, Bosch E. Low serum progesterone on the day of embryo transfer is associated with a diminished ongoing pregnancy rate in oocyte donation cycles after artificial endometrial preparation: a prospective study. Hum Reprod. 2017 Dec 1;32(12):2437-2442. doi: 10.1093/humrep/dex316. PMID 29040638
- [Background] Yovich JL, Conceicao JL, Stanger JD, Hinchliffe PM, Keane KN. Mid-luteal serum progesterone concentrations govern implantation rates for cryopreserved embryo transfers conducted under hormone replacement. Reprod Biomed Online. 2015 Aug;31(2):180-91. doi: 10.1016/j.rbmo.2015.05.005. Epub 2015 May 18. PMID 26099447